CLINICAL TRIAL: NCT03064139
Title: Improving Walking Quality and Quantity in Osteoarthritis (IWALQQ-OA): A Feasibility Study
Brief Title: Improving Walking Quality and Quantity in Osteoarthritis (IWALQQ-OA)
Acronym: IWALQQ-OA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study disrupted due to COVID-19. Interim data analyses in progress.
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Boston University (Other); University of Delaware (Other)
Responsible Party: Principal Investigator, Deepak Kumar, Assistant Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4428E
Record Dates: First submitted 2017-02-14; First posted 2017-02-24 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Knee Osteoarthritis
Keywords: physical activity; gait; biomechanics; mindfulness
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCG - Mindful Walking (Experimental): Participants will be trained in mindful walking technique
  Interventions: Behavioral: MCG
- SCG - Education and Self-Care (Active Comparator): Participants will receive education in self-management of knee OA
  Interventions: Behavioral: SCG

INTERVENTIONS:
Behavioral: MCG — Community-based in person group training n mindful walking over 11 sessions in 6-months+ Activity monitor with feedback on activity levels
  Arms: MCG - Mindful Walking
Behavioral: SCG — Community-based in person group education in management of knee osteoarthritis (importance of physical activity, weight management, etc.) over 11 sessions in 6 months + Activity monitor with feedback on activity levels
  Arms: SCG - Education and Self-Care

SUMMARY:
This study evaluates the feasibility of a mindful walking intervention for management of knee osteoarthritis. Participants will be randomly assigned to receive one of two interventions i.e. mindful walking intervention or a self-care intervention.

DETAILED DESCRIPTION:
People with knee osteoarthritis have low levels of physical activity, especially walking activity. They also walk with abnormal walking biomechanics that are associated with greater knee loading. Therefore, it is important to increase the levels of walking activity in people with knee osteoarthritis, but also change their walking patterns to reduce knee loading.

This study will last 12 months and participants will be randomized into 2 groups. For the first 6-months, half of the participants will attend sessions at a community location that include training in mindful walking technique. The other half will meet for the same frequency and duration at a community location for education on osteoarthritis and its management (focusing on symptom management, importance of physical activity, weight management, etc.). Both groups will also receive a wrist-worn activity monitor and a smartphone application that they will use throughout the study. After 6-months all participants will be allowed to practice on their own.

All participants will complete gait analysis, knee MRI, questionnaires, physical function assessment at baseline and at 6-months. All participants will also complete questionnaires at 3,9, and 12 months. Weekly physical activity and knee pain data will be collected using the mobile health technology for 12- months.

ELIGIBILITY:
Inclusion Criteria:

* age 50-80 years
* BMI ≤40 kg/m2
* Meet American College of Rheumatology clinical and/or clinical+radiographic criteria for knee osteoarthritis
* Knee pain score ≥ 4 during last week
* Predominantly medial knee pain
* Predominantly medial knee radiographic osteoarthritis with or without radiographic patellofemoral osteoarthritis
* Ability to ambulate for a minimum of 20 minutes, without any assistive device
* Available for the study duration
* Own a smartphone
* Can speak and understand English

Exclusion Criteria:

* Contraindications to exercise
* Using orthotics for knee pain such as knee braces, wedge insoles
* Knee injection in previous 3-months
* Currently receiving physical therapy for knee pain
* Planning major treatment for knee pain (e.g., physical therapy, surgery) in next 6 months
* Self-reported joint diseases like rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, gout, etc.
* Self-reported total joint replacement in any lower extremity joint
* Self-reported neurological conditions like stroke, Parkinson's disease, etc.
* Self-reported muscular disease like muscle dystrophy
* Self-reported musculoskeletal or neurologic conditions that affect gait.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Adherence (in %) | 6-months
  Measured as % of in-person training sessions attended by participants
Retention (in %) | 6-months
  Measured as the % of participants returning for the post-intervention assessment

SECONDARY OUTCOMES:
Medial knee contact force during walking (in Newton) | Change from baseline to 6-months
  Medial knee contact force derived using an EMG-Driven musculoskeletal model
Average Daily Activity Count | Change from baseline to 6-months
  Measured using an activity monitor worn by the participants
Knee injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale | Change from baseline to 6-months
  Patient-reported outcome

OTHER OUTCOMES:
Arthritis Self Efficacy Scale (ASES) | Change from baseline to 6-months
  Patient reported outcome
Five Facet Mindfulness Questionnaire (FFMQ) | Change from baseline to 6-months
  Patient reported outcome
Multidimensional Assessment of Interoceptive Awareness (MAIA) questionnaire | Change from baseline to 6-months
  Patient reported outcome
30 second chair stand test (in counts) | Change from baseline to 6-months
  Number of time a participant can stand from a chair
40 meter fast paced walk test (in seconds) | Change from baseline to 6-months
  Time taken to cover 40 meters while walking at a fast pace
Stair Climbing Test (in seconds) | Change from baseline to 6-months
  Time taken to ascend and descend a set of stairs
Knee cartilage composition | Change from baseline to 6-months
  MRI t1rho and t2 relaxation times
Pain sensitization | Change from baseline to 6-months
  Pressure pain threshold, Temporal summation, and conditioned pain modulation

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kumar, PT, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee S, Neogi T, Costello KE, Senderling B, Stefanik JJ, Frey-Law L, Kumar D. Association of mechanical temporal summation of pain with muscle co-contraction during walking in people with knee osteoarthritis. Clin Biomech (Bristol). 2023 Dec;110:106105. doi: 10.1016/j.clinbiomech.2023.106105. Epub 2023 Sep 22. PMID 37778085